CLINICAL TRIAL: NCT07265934
Title: Beneficial Effects of a Food Supplement in Capsule Form and a Functional Chocolate Bar, Both Containing SYNBIO® Probiotic Strains and Grape Marc Plant Extract, on Healthy Adults.
Brief Title: Impact of Supplementation of Probiotics and Grape Marc on Psychological Well-being of Healthy Adults
Acronym: Rescue-bio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synbiotec Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Rescue-bio
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B (Active Comparator): Functional bars administration
  Interventions: Other: Probiotic bars
- Group C (Active Comparator): Dietary supplement administration
  Interventions: Dietary Supplement: Probiotic capsules

INTERVENTIONS:
Other: Probiotic bars — The functional bar contains two probiotic bacterial strains, Lacticaseibacillus rhamnosus IMC 501® and Lacticaseibacillus paracasei IMC 502® at a concentration of 10E9 live cells per gram in a 1:1 combination (SYNBIO, European patent EP 1743042) and 1% grape marc extract; Each participant received one box containing 30 bars, one bar per day for 4 weeks.
  Arms: Group B
Dietary Supplement: Probiotic capsules — The dietary supplement consists of capsules containing two probiotic bacterial strains, Lacticaseibacillus rhamnosus IMC 501® and Lacticaseibacillus paracasei IMC 502® at a concentration of 10E9 live cells per gram in a 1:1 combination (SYNBIO, European patent EP 1743042) and 1% grape marc extract. Each participant received one bottle containing 30 capsules, one capsule per day for 4 weeks.
  Arms: Group C

SUMMARY:
An open-label, baseline-controlled (pre-post) pilot study to assess the maintenance and/or improvement of both physical and mental well-being in subjects who daily consume either a food supplement or a functional food containing both the SYNBIO® probiotic blend and the dry grape marc extract. A target number of 40 healthy individuals will be recruited who meet the inclusion and exclusion criteria, who will be assessed upon enrollment and who have signed informed consent. Subjects will be randomly assigned to either the functional food or dietary supplement groups.

DETAILED DESCRIPTION:
The present clinical trial is a pilot open label, baseline-controlled (pre/post) experimental study, with a, a 2-week run-in period, 4-week intervention period and a further 2-week follow-up period without intervention to evaluate the potential prolonged effect of the functional products. Specifically, the supplementation should improve the parameters related to physical and mental well-being of subjects. Healthy adult participants were recruited and randomized into two treatment groups in a 1:1 ratio. Subjects will be randomly assigned to either the functional food or dietary supplement groups. The study will consist of three meetings at the coordinating center. The first visit will be for enrollment. Through an interview, the investigator will verify that the volunteer meets the inclusion criteria. The volunteer will receive an informed consent form to sign and the study protocol information sheet, which explains the study's progress in a simple and clear manner. The investigator will answer any questions and concerns the volunteer may have regarding the study. Subjects will be randomly assigned to either the functional food or dietary supplement group. Recruited subjects will be given questionnaires to complete independently. The second meeting will take place at the end of the month of taking the study products and will consist of the administration of the end-of-treatment questionnaires. The third and final meeting, two weeks after the end of treatment, will involve completing the questionnaires again to assess the possible persistence of the benefits that taking the products may have produced.

ELIGIBILITY:
Inclusion Criteria:

* men and women between 18 and 55 years;
* healthy based on medical history;
* commitment to comply with all study procedures;
* have a moderate level of stress (score 13-20) based on the Cohen Perceived Stress Scale (PSS-10);
* signing of informed consent.

Exclusion Criteria:

* significant acute or chronic illnesses and/or an immunocompromised state
* pregnant women who are breastfeeding or planning to become pregnant during the study period
* subjects with clinically significant gastrointestinal tract disease, subjects with allergy or sensitivity to the active or inactive ingredients of the investigational product
* subjects who had used antibiotics in the month prior to enrolment or who had used probiotics continuously in the two months prior to enrolment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress levels | After 4 weeks consumption of the study product
  to evaluate the effect of the probiotic products on perceived stress levels measured using the Perceived Stress Scale (PSS). 5-point scale from 0 (never) to 4 (very often).

SECONDARY OUTCOMES:
Assessment of sleep quality | After 4 week consumption of the study product
  To evaluate the sleep quality through the PSQI (Pittsburgh Sleep Quality Index) 4 weeks after consumption of the study product. 0-3 interval scale , global PSQI score (range 0-21), the lower the PSQI global score, the better the sleep quality.
Assessment of sleep quality | After 2 weeks follow-up (week 6)
  To evaluate the sleep quality through the PSQI (Pittsburgh Sleep Quality Index) 2 weeks after the end of the study product consumption period. 0-3 interval scale , global PSQI score (range 0-21), the lower the PSQI global score, the better the sleep quality.
Assessment of physical activity | After 4 weeks consumption of study product
  To evaluate the physical activity through the IPAQ (International Physical Activity Questionnaire) 4 week after consumption of the study product
Assessment of physical activity | After 2 weeks follow-up (week 6)
  To evaluate physical activity through the IPAQ (International Physical Activity Questionnaire) 2 weeks after the end of the study product consumption period
Changes on health-related quality of life | After 4 weeks consumption of the study product
  To evaluate changes on health-related quality of life through the GIQLI questionnaire 4 weeks after consumption of the study product. Scale from 0 to 4, a global score can be estimated that goes from 0 to 144. The higher the score, the better the result.
Changes on health-related quality of life | After 2 weeks follow-up (week 6)
  To evaluate changes on health-related quality of life through the GIQLI questionnaire 2 weeks after the end of the study product consumption period. Scale from 0 to 4, a global score can be estimated that goes from 0 to 144. The higher the score, the better the result.
Changes in quality of life | After 4 weeks consumption of the study product
  To evaluate changes in quality of life, assessed through the PGWBI questionnaire (The Psychologi-cal General Well-Being Index) 4 weeks after consumption of the study product. Score from 0 (severe stress) to 110 (well-being).
Changes in quality of life | After 2 weeks follow-up (week 6)
  To evaluate changes in quality of life, assessed through the PGWBI questionnaire (The Psychologi-cal General Well-Being Index) 2 weeks after the end of the study product consumption period. Score from 0 (severe stress) to 110 (well-being).
Changes in intestinal function | After 4 weeks consumption of the study product
  To evaluate changes in intestinal function assessed according to the Bristol Stool Form Scale 4 weeks after consumption of the study product
Changes in intestinal function | After 2 weeks follow-up (week 6)
  To evaluate changes in intestinal function assessed according to the Bristol Stool Form Scale 2 weeks after the end of the study product consumption period
Changes in gastrointestinal symptoms | After 4 weeks consumption of the study product
  To evaluate changes in gastrointestinal symptoms assessed through the GSRS questionnaire (Gastrointestinal Symptom Rating Scale) 4 weeks after consumption of the study product. Seven-point Likert scale, from no discomfort (score 1) to very severe discomfort (score 7).
Changes in gastrointestinal symptoms | After 2 weeks follow-up (week 6)
  To evaluate changes in gastrointestinal symptoms assessed through the GSRS questionnaire (Gastrointestinal Symptom Rating Scale) 2 weeks after the end of the study product consumption period. Seven-point Likert scale, from no discomfort (score 1) to very severe discomfort (score 7).
Change in perceived stress levels | After 2 weeks follow-up (week 6)
  To evaluate perceived stress levels measured using the Perceived Stress Scale (PSS) 2 weeks after the end of the study product consumption period. 5-point scale from 0 (never) to 4 (very often).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Verdenelli, Principal Investigator — Synbiotec Srl
Locations (1):
- Centro Universitario Sportivo, University of Camerino, Camerino, Macerata, Italy